CLINICAL TRIAL: NCT03507166
Title: A Multicenter, Open Label，Single Arm，Phase II Study to Evaluate the Effect and Safety of Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection in Subjects With HER2 Positive Metastatic or Unresectable Urothelial Cancer
Brief Title: A Phase II Study of RC48-ADC in Subjects With HER2 Positive Metastatic or Unresectable Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C005
Record Dates: First submitted 2018-04-08; First posted 2018-04-24 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Urothelial Carcinoma; Advanced Cancer
Keywords: RC48-ADC; HER2
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Drug: RC48-ADC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC (Experimental): Participants will receive RC48-ADC every 2 weeks (Q2W) until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: RC48-ADC

INTERVENTIONS:
Drug: RC48-ADC — 2 mg/kg IV every 2 weeks
  Other Names: Recombinant Humanized anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection

SUMMARY:
This study will evaluate the efficacy and safety of intravenous RC48-ADC in patients with local advanced or metastatic HER2 positive endothelial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Male or female, Age ≥ 18 years and < 80 years.
* Predicted survival ≥ 12 weeks.
* Have histologically or cytologically-confirmed diagnosis of inoperable, locally advanced or metastatic urothelial cancer of the bladder, renal pelvis, ureter.
* Have had progression or intolerance following receipt of at least one systemic chemotherapy for advanced or metastatic disease.
* Measurable disease according to RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* HER2-positive status confirmed by the central laboratory: IHC 2+ or 3+; Subject is able to provide specimens from primary or metastatic lesions for HER2 tests
* Adequate organ function, evidenced by the following laboratory results:

Cardiac ejection fraction ≥ 50 %. Hemoglobin ≥ 9g/dL; Absolute neutrophil count ≥ 1.5×109 /L Platelets ≥ 100×109 /L; Total bilirubin ≤ 1.5× ULN; Without liver metastasis: ALT and AST ≤ 2.5 x ULN; With liver metastasis: ALT and AST ≤ 5 x ULN; Serum creatinine ≤1.5×ULN or creatinine clearance (CrCl) ≥ 50 mL/min as calculated by the Cockcroft-Gault equation.

* All female subjects will be considered to be of child-bearing potential unless they are postmenopausal, or have been sterilized surgically.Female subjects of child-bearing potential must agree to use two forms of highly effective contraception. Male subjects and their female partner who are of child-bearing potential must agree to use two forms of highly effective contraception.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Known hypersensitivity to Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection.
* History of receiving any anti-cancer drug/biologic treatment within 4 weeks prior to trial treatment.
* History of receiving Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection.
* History of major surgery within 4 weeks of planned start of trial treatment.
* Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
* Currently known active infection with HIV or tuberculosis.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
* known central nervous system metastases.
* Pregnancy or lactation.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate （ORR） | up to 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
ORR of HER2-positive patients | up to 24 months
  Tumor response was assessed by investigator according to RECIST v1.1
Progression Free Survival (PFS) | up to 24 months
  Tumor response was assessed by investigator according to RECIST v1.1
Duration of Response (DOR) | up to 24 months
  DOR was defined as the time from first documented OR to first documented PD or death from any cause, whichever occurred earlier
Disease control rate (DCR) | up to 24 months
  DCR was defined as the proportion of patients who achieved an objective response or maintained stable disease during the study
Overall Survival(OS) | up to 24 months
  OS was defined as the time from the first study treatment to the date of death from any cause
Adverse Events | 28 days after the last dose of study treatment
  Incidence of Adverse Events

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, N/A = Not Applicable
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, N/A = Not Applicable

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheng X, Wang L, He Z, Shi Y, Luo H, Han W, Yao X, Shi B, Liu J, Hu C, Liu Z, Guo H, Yu G, Ji Z, Ying J, Ling Y, Yu S, Hu Y, Guo J, Fang J, Zhou A, Guo J. Efficacy and Safety of Disitamab Vedotin in Patients With Human Epidermal Growth Factor Receptor 2-Positive Locally Advanced or Metastatic Urothelial Carcinoma: A Combined Analysis of Two Phase II Clinical Trials. J Clin Oncol. 2024 Apr 20;42(12):1391-1402. doi: 10.1200/JCO.22.02912. Epub 2023 Nov 21. PMID 37988648
- [Derived] Sheng X, Yan X, Wang L, Shi Y, Yao X, Luo H, Shi B, Liu J, He Z, Yu G, Ying J, Han W, Hu C, Ling Y, Chi Z, Cui C, Si L, Fang J, Zhou A, Guo J. Open-label, Multicenter, Phase II Study of RC48-ADC, a HER2-Targeting Antibody-Drug Conjugate, in Patients with Locally Advanced or Metastatic Urothelial Carcinoma. Clin Cancer Res. 2021 Jan 1;27(1):43-51. doi: 10.1158/1078-0432.CCR-20-2488. Epub 2020 Oct 27. PMID 33109737